CLINICAL TRIAL: NCT02900742
Title: Study of Chinese Medicine Plus Chemotherapy Maintenance Versus Chemotherapy Maintenance in Advanced Non Small Cell Lung Cancer: A Randomized Double-blind Controlled Clinical Trial
Brief Title: Clinical Study of Chinese Medicine Plus Chemotherapy Maintenance in Advanced Non Small Cell Lung Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shanghai University of Traditional Chinese Medicine (Other)
Collaborators: Shanghai Chest Hospital (Other); Shanghai Pulmonary Hospital, Shanghai, China (Other)
Responsible Party: Principal Investigator, Ling Xu, Principal Investigator, Shanghai University of Traditional Chinese Medicine
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LH128
Record Dates: First submitted 2016-07-25; First posted 2016-09-14 (Estimated); Last update posted 2019-04-12 (Actual); Status verified 2019-04

CONDITIONS: Cancer
Keywords: lung cancer; traditional Chinese medicine; maintenance therapy; chemotherapy
MeSH Terms: conditions — Neoplasms; Lung Neoplasms | interventions — Gemcitabine; Pemetrexed; Docetaxel

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- TCM granules plus Chemotherapy (Experimental): TCM granules: oral granules, "YiQiFang" or "YangYinFang" or "YiQiYangYinFang", four packages, twice a day until progression or unacceptable toxicity; Chemotherapy: Gemcitabine® 1250 mg/㎡, ivgtt 30 min,days 1,8,every 21 days or Pemetrexed® 500 mg/㎡, ivgtt 30 min, day 1, every 21 days or Docetaxel® 75 mg/㎡, ivgtt 30 min, day 1, every 21 days until progression or unacceptable toxicity.
  Interventions: Drug: YiQiFang; Drug: YangYinFang; Drug: YiQiYangYinFang; Drug: Gemcitabine®; Drug: Pemetrexed®; Drug: Docetaxel®
- Placebo granules plus Chemotherapy (Placebo Comparator): Placebo granules: oral granules, oral granules, which the taste and smell are similar to experimental TCM granules and has no therapeutic effect, four packages, twice a day; Chemotherapy: Gemcitabine® 1250 mg/㎡, ivgtt 30 min,days 1,8,every 21 days or Pemetrexed® 500 mg/㎡, ivgtt 30 min, day 1, every 21 days or Docetaxel® 75 mg/㎡, ivgtt 30 min, day 1, every 21 days until progression or unacceptable toxicity.
  Interventions: Drug: Gemcitabine®; Drug: Pemetrexed®; Drug: Docetaxel®; Drug: placebo granules

INTERVENTIONS:
Drug: YiQiFang — Prescriptions formulated into TCM granules origin from Professor Liu Jia-xiang in Longhua hospital. Package of granules is made into three types with functions such as benefiting Qi, benefiting Yin and detoxication recipe. YiQiFang: Patients with Qi deficiency syndrome are administered two packages of each benefiting Qi and detoxication recipe, four packages, twice a day, until progression or unacceptable.
  Arms: TCM granules plus Chemotherapy
Drug: YangYinFang — Prescriptions formulated into TCM granules origin from Professor Liu Jia-xiang in Longhua hospital. Package of granules is made into three types with functions such as benefiting Qi, benefiting Yin and detoxication recipe. YangYinFang: Patients with Yin deficiency syndrome are administered two packages of each benefiting Yin and detoxication recipe, four packages, twice a day, until progression or unacceptable.
  Arms: TCM granules plus Chemotherapy
Drug: YiQiYangYinFang — Prescriptions formulated into TCM granules origin from Professor Liu Jia-xiang in Longhua hospital. Package of granules is made into three types with functions such as benefiting Qi, benefiting Yin and detoxication recipe. YiQiYangYinFang: Patients with Qi and Yin deficiency syndrome are administered one package of each benefiting Qi and benefiting Yin and two packages of detoxication recipe, four packages, twice a day, until progression or unacceptable.
  Arms: TCM granules plus Chemotherapy
Drug: Gemcitabine® — "Gemcitabinie®","Gemzar",1250 mg/㎡, ivgtt 30 min,days 1,8,every 21 days until progression or unacceptable toxicity develops.
  Other Names: Gemzar
Drug: Pemetrexed® — "Pemetrexed®","Alimta",500 mg/㎡, ivgtt 30 min, day 1, every 21 days until progression or unacceptable toxicity develops.
  Other Names: Alimta
Drug: Docetaxel® — "Docetaxel®","Taxotere",75 mg/㎡, ivgtt 30 min, day 1, every 21 days until progression or unacceptable toxicity.
  Other Names: Taxotere
Drug: placebo granules — Oral granules, which the taste and smell are similar to experimental TCM granules, has no therapeutic effect, four packages, twice a day, until progression or unacceptable.
  Arms: Placebo granules plus Chemotherapy

SUMMARY:
The investigators performed a randomized, prospective study method on observation of Traditional Chinese Medicine(TCM) combined with chemotherapy maintenance to prolong the efficacy of long-term survival of advanced non small cell lung cancer(NSCLC) patients.The investigators plan to involve 100 cases for observation in 3 years (50 cases for chemotherapy maintenance, 50 cases for chemotherapy maintenance plus TCM), expecting that integrated TCM combined with chemotherapy maintenance has a better efficacy on prolonging progression-free survival time, overall survival, improving quality of life(QOL) of patients than that of chemotherapy maintenance.

DETAILED DESCRIPTION:
Maintenance therapy refers to systemic therapy that may be given for patients with advanced NSCLC after 4 to 6 cycles of first-line chemotherapy. However, patients are only candidates for maintenance therapy if they have responded to their previous treatment or have stable disease and their tumors have not progressed. Pemetrexed, docetaxel and gemcitabine have been approved for chemotherapy maintenance in the NCCN Guide. Chemotherapy maintenance can be partly extend patient's TTP, but the toxicity and the side effects of chemotherapy will decrease the QOL, and even lose the opportunity to receive subsequent therapy. Besides, high cost of chemotherapy will cause greater economic pressure on patients. Our preliminary studies have shown that traditional Chinese medicine (TCM) can prolong survival time and improve QOL, but high-level evidences are needed.

The investigators perform a multicenter, randomized, double-blind controlled, prospective study in advanced non small cell lung cancer patients with stage Ⅲ～Ⅳ.Advanced NSCLC patients after first-line chemotherapy will choose maintenance therapy according to the patient's wishes, including targeted therapy maintenance, chemotherapy maintenance and maintenance of TCM therapy. Patients who choose chemotherapy maintenance are randomized over observational group (TCM granules plus chemotherapy maintenance),and control group (TCM placebo plus chemotherapy maintenance). The treatment should be continued until evidence of disease progression or unacceptable toxicity, and after that regular follow-up will be arranged. The primary efficacy assessments are: PFS (progression-free survival）; Secondary efficacy assessments are: (1) OS(overall survival); (2) Objective response rate; (3) TTP（Time-to-Progression）; (4) QOL (Functional Assessment of Cancer therapy-lung, FACT-L4.0 scales;Lung Cancer Symptom Scale,LCSS); (5)other efficacy assessments are: 1) TCM symptoms changes; 2) Toxicity, side effects and security of the treatments will be assessed at the same time.The investigators expect that integrated TCM combined with chemotherapy maintenance has a better efficacy on prolonging progression-free survival time, overall survival, improving QOL of patients than that of chemotherapy maintenance. Therefore our study can provide evidences for optimizing and promoting integrated TCM combined with Western Medicine treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Pathologically or cytologically confirmed of stage IIIa-IV NSCLC;
2. The efficacy evaluation of the first-line therapy is progression-free including complete response(CR), partial response(PR) and stable disease(SD);
3. At the age of 18 -75 years old;
4. Physical status score (ECOG PS) ≤ 2 scores;
5. Estimated life expectancy of at least 12 weeks;
6. Participants have no major organ dysfunction: hemoglobin ≥10 g/dL, absolute neutrophil count (ANC) ≥1.5*109/L, platelets ≥100 *109/L,bilirubin ≤1.5ULN, alkaline phosphatase (AP), aspartate transaminase (AST) and alanine transaminase (ALT) ≤2.5 upper limited number(ULN) (AP, AST, ALT ≤5ULN is acceptable if liver has tumor involvement).INR≤1.5, APTT in the normal range( 1.2DLN-1.2ULN),creatinine ≤1.5ULN;
7. Planning for chemotherapy maintenance.
8. Informed consent from the patient.

Exclusion Criteria:

1. The efficacy evaluation of the first-line therapy is progressive disease;
2. Patient with other malignant tumor except NSCLC 5 years previous to study entry;
3. Patient already receiving targeted therapy or other anticancer treatment;
4. Allergic to chemotherapy drugs;
5. Estimated life expectancy less than 12 weeks;
6. History of cardiovascular disease: Congestive Heart Failure > grade II in NYHA.Unstable angina patients (have angina symptoms in rest) or a new occurrence of angina (began in the last 3 months) or myocardial infarction happens in the last 6 months;
7. Pregnant or child breast feeding women;
8. Mental or cognitive disorders.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2013-03; Primary Completion 2016-12-30 (Actual); Study Completion 2017-06-01 (Actual)

PRIMARY OUTCOMES:
Overall survival(OS) | 2 months
  It referred to the interval time from the first date of randomization to that of death for any reason, the end of the study, or loss of follow-up.

SECONDARY OUTCOMES:
Progression-free survival(PFS) | 2 months
  Time from start of the study treatment to date of objective tumour progression (excluding clinical deterioration without evidence of objective progression).
Overall response rate(ORR) | 2 months
  The ORR (complete response (CR) plus partial response (PR)) was determined by the Response Evaluation Criteria In Solid Tumors (RECIST) (Eisenhauer et al, 2009) version 1.1.in Solid Tumors (RECIST1.1).
Quality of life (QOL) | 2 months
  QOL is assessed using Functional Assessment of Cancer therapy-lung (FACT-L) questionnaire .
Quality of life(QOL) | 2 months
  QOL was assessed using Functional Assessment of Cancer therapy-lung(FACT-L) and Lung Cancer Symptom Scale(LCS).

OTHER OUTCOMES:
TCM symptoms changes | 2 months
  TCM symptoms changes are according to the lung cancer symptom classification quantization table in "Guiding Principles for Clinical Research of Traditional Chinese Medicine in the Treatment of Lung Cancer (2002 Edition)".
Safety assessment evaluated according to Common Toxicity Criteria | 2 months
  Safety assessment is evaluated according to Common Toxicity Criteria (CTC 3.0).

CONTACTS AND LOCATIONS:
Overall Officials: Ling Xu, MD & PhD, Principal Investigator — Longhua Hospital Affiliated to Shanghai University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wang Q, Jiao L, Wang S, Chen P, Bi L, Zhou D, Yao J, Li J, Chen Z, Jia Y, Zhang Z, Shen W, Zhu W, Xu J, Gao Y, Gong Y, Xu L. Maintenance Chemotherapy With Chinese Herb Medicine Formulas vs. With Placebo in Patients With Advanced Non-small Cell Lung Cancer After First-Line Chemotherapy: A Multicenter, Randomized, Double-Blind Trial. Front Pharmacol. 2018 Nov 6;9:1233. doi: 10.3389/fphar.2018.01233. eCollection 2018. PMID 30459612
- See also: full paper — https://www.frontiersin.org/articles/10.3389/fphar.2018.01233/full